CLINICAL TRIAL: NCT02520141
Title: A Phase II Study of Ramucirumab for Advanced, Pre-Treated Biliary Cancers
Brief Title: Ramucirumab in Treating Patients With Advanced or Metastatic, Previously Treated Biliary Cancers That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0393; NCI-2015-01442 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0393 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-08-05; First posted 2015-08-11 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Cholangiocarcinoma; Liver and Intrahepatic Bile Duct Carcinoma; Stage III Gallbladder Cancer AJCC v7; Stage III Intrahepatic Cholangiocarcinoma AJCC v7; Stage IIIA Gallbladder Cancer AJCC v7; Stage IIIB Gallbladder Cancer AJCC v7; Stage IV Gallbladder Cancer AJCC v7; Stage IVA Gallbladder Cancer AJCC v7; Stage IVA Intrahepatic Cholangiocarcinoma AJCC v7; Stage IVB Gallbladder Cancer AJCC v7; Stage IVB Intrahepatic Cholangiocarcinoma AJCC v7; Unresectable Gallbladder Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Carcinoma, Hepatocellular; Gallbladder Neoplasms | interventions — Ramucirumab

ARMS (1):
- Treatment (ramucirumab) (Experimental): Patients receive ramucirumab IV over 60 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Ramucirumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Ramucirumab — Given IV
  Other Names: anti-VEGFR-2 fully human monoclonal antibody IMC-1121B; Cyramza; IMC-1121B; LY3009806; Monoclonal Antibody HGS-ETR2

SUMMARY:
This phase II trial studies how well ramucirumab works in treating patients with previously treated biliary cancers that have spread to other places in the body and usually cannot be cured or controlled with treatment (advanced) or have spread to other places in the body (metastatic) and cannot be removed by surgery. Immunotherapy with monoclonal antibodies, such as ramucirumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the progression-free survival (PFS) of ramucirumab in advanced biliary cancers (intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, and gallbladder cancer) who have received prior chemotherapy.

SECONDARY OBJECTIVES:

I. Determine the response rate (RR) and disease control rate (partial response + complete response + stable disease) of ramucirumab in advanced biliary cancers.

II. Determine overall survival (OS) of ramucirumab in advanced biliary cancers. III. Evaluate the toxicity of ramucirumab in advanced biliary cancers.

EXPLORATORY OBJECTIVES:

I. Correlate the carbohydrate antigen (CA) 19-9 response (defined as > 50% decrease from baseline) with tumor response, PFS and OS.

II. Correlate baseline tumor gene expression profile with PFS. III. Correlate pre- and post-therapy computed tomography (CT) imaging to quantify iodine content, atomic numbers, and Z-values and correlate with response.

OUTLINE:

Patients receive ramucirumab intravenously (IV) over 60 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have cholangiocarcinoma, gallbladder cancer or adenocarcinoma on liver biopsy with clinical features consistent with biliary primary/cholangiocarcinoma
* Metastatic or unresectable disease documented on diagnostic imaging studies
* Must have received at least one regimen containing gemcitabine chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Total bilirubin =< 1.5 mg/dL (25.65 mol/L)
* Aspartate transaminase (AST) and alanine transaminase (ALT) =< 3.0 times the upper limit of normal ([ULN]; or 5.0 times the ULN in the setting of liver metastases)
* Absolute neutrophil count (ANC) >= 1000/uL
* Hemoglobin >= 9 g/dL (5.58 mmol/L)
* Platelets >= 100,000/uL
* The patient does not have:

  * Cirrhosis at a level of Child-Pugh B (or worse) or
  * Cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis; clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis
* Serum creatinine =< 1.5 times the ULN or
* Creatinine clearance (measured via 24-hour urine collection) >= 40 mL/minute (that is, if serum creatinine is > 1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed
* The patient's urinary protein is =< 1 positive (+) (=< 30-100 mg/dl) on dipstick or routine urinalysis (urinary analysis [UA]; if urine dipstick or routine analysis is >= 2+ (>=100-300 mg/dl), a 24-hour urine collection for protein must demonstrate < 1000 mg of protein in 24 hours to allow participation in this protocol)
* The patient must have adequate coagulation function as defined by international normalized ratio (INR) =< 1.5 and
* Partial thromboplastin time (PTT) (PTT/activated partial thromboplastin time [aPTT]) < 1.5 x ULN)
* Patients on full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin; if receiving warfarin, the patient must have an INR =< 3.0 and no active bleeding (that is, no bleeding within 14 days prior to first dose of protocol therapy) or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices)
* The patient, if sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods)
* Female patients of childbearing potential must have a negative serum pregnancy test within 7 days
* Patients must sign an informed consent and authorization indicating that they are aware of the investigational nature of this study and the known risks involved
* In the ten patient expanded cohort, patients diagnosed with deoxyribonucleic acid (DNA) repair or FGFR genetic aberrations will be enrolled

Exclusion Criteria:

* The patient has experienced any grade 3-4 gastrointestinal (GI) bleeding within 3 months prior to enrollment
* Prior therapy with any agent targeting the vascular endothelial growth factor receptor (VEGFR) pathway to include bevacizumab, pazopanib, and other anti-angiogenesis inhibitors
* The patient has a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism, including portal venous thrombosis (venous port or catheter thrombosis, incidental pulmonary embolism diagnosed on imaging studies or superficial venous thrombosis are not considered significant) during the 3 months prior to randomization
* The patient has experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to enrollment
* The patient has uncontrolled or poorly-controlled hypertension (> 160 mmHg systolic or > 100 mmHg diastolic for > 4 weeks) despite standard medical management
* The patient has a serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment
* The patient has undergone major surgery within 28 days prior to enrollment, or subcutaneous venous access device placement within 7 days prior to enrollment
* The patient is receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs ([NSAIDs], including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents; once-daily aspirin use (maximum dose 325 mg/day) is permitted
* The patient has elective or planned major surgery to be performed during the course of the clinical trial
* The patient is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachna T Shroff, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: MD Anderson Cancer Center Houston Tx
Groups:
- Phase II Open-label, Single Arm Study of Ramucirumab Administered at 8 mg/kg IV.: Phase II, single-arm trial for advanced, unresectable, pre-treated patients with BTC. Eligible patients received ramucirumab 8 mg/kg IV on day 1 of a 14-day cycle until progression or intolerable toxicity.
Period: Overall Study
Arm/Group | Phase II Open-label, Single Arm Study of Ramucirumab Administered at 8 mg/kg IV.
Started | 61
Completed | 60
Not Completed | 1
Not completed — Rapid decline clinically and thus unable to enroll | 1

BASELINE CHARACTERISTICS:
Arm/Group | Phase II Open-label, Single Arm Study of Ramucirumab Administered at 8 mg/kg IV.
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 58.5 [41 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race and Ethnicity Not Collected
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race and Ethnicity Not Collected
Region of Enrollment [Count of Participants; unit: Participants] — Region of Enrollment data not collected Population: Region of Enrollment data not collected

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival of Ramucirumab in Advanced Biliary Cancers
Description: Progression free survival is measured using 95% confidence intervals. From the date of treatment start to the date of disease progression or to the date of death, whichever occurs first, or to the last follow-up date if patients are alive without disease progression, assessed up to at least 3 months post-treatment
Time Frame: Up to 6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II Open-label, Single Arm Study of Ramucirumab Administered at 8 mg/kg IV.
Number analyzed (Participants) | 60
months | 3.2 [2.1 to 4.8]

2. Secondary Outcome: Overall Survival (OS)
Description: Overal Survival (OS): the time from treatment initiation to death from any cause. OS functions were estimated using the Kaplan-Meier method .
Time Frame: Up to 6 years
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase II Open-label, Single Arm Study of Ramucirumab Administered at 8 mg/kg IV.: Phase II, single-arm trial for advanced, unresectable, pre-treated patients with BTC with ECOG 0/1, adequate liver, renal, and marrow functions
Arm/Group | Phase II Open-label, Single Arm Study of Ramucirumab Administered at 8 mg/kg IV.
Number analyzed (Participants) | 60
Months | 9.5 [5.81 to 13.6]

3. Secondary Outcome: Overall Response Rate (RR)
Description: The proportion of patients with the best overall response of complete response or partial response (PR)]
Time Frame: Up to 6 years
Measure: Number; unit: participants
Arm/Group | Phase II Open-label, Single Arm Study of Ramucirumab Administered at 8 mg/kg IV
Number analyzed (Participants) | 60
participants | 1

4. Secondary Outcome: Percentage of Disease Control Rate
Description: Partial Response + Complete Response + Stable Disease (ORR + Stable Disease)
Time Frame: Up to 6 years
Measure: Number; unit: percentage
Arm/Group | Phase II Open-label, Single Arm Study of Ramucirumab Administered at 8 mg/kg IV
Number analyzed (Participants) | 60
percentage | 45

ADVERSE EVENTS:
Time Frame: Up to 6 years
Description: NCI CTCAE version 4.0.
Arm/Group | Phase II Open-label, Single Arm Study of Ramucirumab Administered at 8 mg/kg IV.
All-Cause Mortality (participants affected / at risk) | 60/60
Serious Adverse Events (participants affected / at risk) | 1/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II Open-label, Single Arm Study of Ramucirumab Administered at 8 mg/kg IV. (N=60)
Upper GI Bleeding (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase II Open-label, Single Arm Study of Ramucirumab Administered at 8 mg/kg IV. (N=60)
Proteinuria (Investigations) | 23
Thrombocytopenia (Investigations) | 13
Anemia (Investigations) | 11
Hyperbilirubinemia (Investigations) | 9
Alkaline phosphatase increase (Investigations) | 9
AST increase (Investigations) | 9
Hyponatremia (Investigations) | 9
ALT increase (Investigations) | 8
Hyperkalemia (Investigations) | 7
Hypercalcemia (Investigations) | 5
Hypomagnesemia (Investigations) | 5
Creatinine (Investigations) | 4
Hypoalbuminemia (Investigations) | 3
Hematuria (Investigations) | 2
Hypermagnesemia (Investigations) | 2
Hypoglycemia (Investigations) | 2
Hypokalemia (Investigations) | 2
Prolonged PTT (Investigations) | 1
Hyperglycemia (Investigations) | 1
Hypocalcemia (Investigations) | 1
Hypophosphatemia (Investigations) | 1
Hypotension (Investigations) | 1
Increased INR (Investigations) | 1
Hypertension (Vascular disorders) | 25
Upper GI hemorrhage (Gastrointestinal disorders) | 1
Pulmonary embolism (Vascular disorders) | 1
Fatigue (General disorders) | 23
Headache (Nervous system disorders) | 21
Nausea and vomiting (Gastrointestinal disorders) | 16
Abdominal pain (Gastrointestinal disorders) | 14
Diarrhea (Gastrointestinal disorders) | 14
Lower extremity edema (Vascular disorders) | 13
Anorexia (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 11
Fever (General disorders) | 11
Dizziness (Nervous system disorders) | 9
Ascites (Gastrointestinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Extremity pain (Nervous system disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 6
Urinary tract infection (Renal and urinary disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Neuropathy (Nervous system disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 4
Allergic rhinitis (Immune system disorders) | 4
Chest pain (Respiratory, thoracic and mediastinal disorders) | 4
Diaphoresis (General disorders) | 4
Mucositis (Gastrointestinal disorders) | 4
Sepsis (Infections and infestations) | 4
Confusion (Nervous system disorders) | 3
Dehydration (General disorders) | 3
Gastric obstruction (Gastrointestinal disorders) | 3
Gastroesophageal reﬂux (Gastrointestinal disorders) | 3
Skin rash (Skin and subcutaneous tissue disorders) | 3
Chills (General disorders) | 2
Cholangitis (Gastrointestinal disorders) | 2
Hot ﬂashes (General disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (General disorders) | 2
Thrombocytopenic purpura (Vascular disorders) | 2
Biliary obstruction (Gastrointestinal disorders) | 1
Blurry vision (Nervous system disorders) | 1
Delirium (Nervous system disorders) | 1
Facial edema (General disorders) | 1
Epistaxis (Vascular disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastroparesis (Gastrointestinal disorders) | 1
Hiccups (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT02520141/Prot_SAP_000.pdf